CLINICAL TRIAL: NCT04255017
Title: An Open, Prospective/Retrospective, Randomized Controlled Cohort Study to Compare the Efficacy of Three Antiviral Drugs(Abidol Hydrochloride, Oseltamivir and Lopinavir/Ritonavir) in the Treatment of 2019-nCoV Pneumonia.
Brief Title: A Prospective/Retrospective,Randomized Controlled Clinical Study of Antiviral Therapy in the 2019-nCoV Pneumonia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ20200128
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: 2019-nCoV
MeSH Terms: interventions — Oseltamivir; Lopinavir

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Symptomatic supportive treatment (No Intervention): Symptomatic supportive treatment
- Abidol hydrochloride was added on the basis of group I. (Experimental): Abidol hydrochloride 0.2g once,3 times a day,2 weeks
  Interventions: Drug: Abidol hydrochloride
- Oseltamivir was added on the basis of group I. (Experimental): Oseltamivir 75mg once,twice a day,2 weeks
  Interventions: Drug: Oseltamivir
- Lopinavir/ritonavir was added on the basis of group I. (Experimental): Lopinavir/ritonavir 500mg once,twice a day,2 weeks
  Interventions: Drug: Lopinavir/ritonavir

INTERVENTIONS:
Drug: Abidol hydrochloride — Abidol hydrochloride (0.2g once, 3 times a day,2 weeks)was added on the basis of group I.
  Arms: Abidol hydrochloride was added on the basis of group I.
Drug: Oseltamivir — Oseltamivir(75mg once, twice a day,2 weeks) was added on the basis of group I.
  Arms: Oseltamivir was added on the basis of group I.
Drug: Lopinavir/ritonavir — Lopinavir/ritonavir (500mg once, twice a day,2 weeks)was added on the basis of group I.
  Arms: Lopinavir/ritonavir was added on the basis of group I.

SUMMARY:
At present, there is no specific and effective antiviral therapy.In this study, an open, prospective/retrospective, randomized controlled cohort study was designed to compare the efficacy of three antiviral drugs in the treatment of 2019-nCoV pneumonia by studying the efficacy of abidol hydrochloride, oseltamivir and lopinavir/ritonavir in the treatment of 2019-nCoV viral pneumonia, and to explore effective antiviral drugs for new coronavirus. To provide reliable evidence-based medicine basis for the treatment of viral pneumonia caused by new coronavirus infection.

ELIGIBILITY:
Inclusion Criteria:

1. 2019-nCoV nucleic acid test was positive.
2. CT of the lung conformed to the manifestation of viral pneumonia.

Exclusion Criteria:

1. Patients who meet any of the contraindications in the experimental drug labeling
2. Patients who do not want to participate in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of disease remission | two weeks
  A: For mild patients : fever, cough and other symptoms relieved with improved lung CT; B:For severe patients : fever, cough and other symptoms relieved with improved lung CT,SPO2> 93% or PaO2/FiO2>300mmHg (1mmHg=0.133Kpa);
Time for lung recovery | two weeks
  Compare the average time of lung imaging recovery after 2 weeks of treatment in each group.

SECONDARY OUTCOMES:
Rate of no fever | two weeks
Rate of respiratory symptom remission | two weeks
Rate of lung imaging recovery | two weeks
Rate of CRP,ES,Biochemical criterion(CK,ALT,Mb) recovery | two weeks
Rate of undetectable viral RNA | two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department and Institute of Infectious Disease, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided